CLINICAL TRIAL: NCT00252317
Title: Acute Haemodynamic Effects of Treatment With ACE-Inhibitors in Patients With Symptomatic Aortic Stenosis (ACCESS)
Brief Title: Acute Haemodynamic Effects of Treatment With Angiotensin Converting Enzyme (ACE)-Inhibitors in Patients With Symptomatic Aortic Stenosis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3d
Record Dates: First submitted 2005-11-10; First posted 2005-11-11 (Estimated); Last update posted 2008-09-03 (Estimated); Status verified 2007-11

CONDITIONS: Aortic Stenosis
Keywords: Aortic stenosis; ACE-inhibitores
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Captopril; trandolapril

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Captopril test dose and Trandolapril
  Interventions: Drug: Captopril and Trandolapril; Drug: Captopril Test Dose and Trandolapril
- 2 (Placebo Comparator)
  Interventions: Drug: Captopril and Trandolapril; Drug: Captopril Test Dose and Trandolapril

INTERVENTIONS:
Drug: Captopril and Trandolapril — Caps Captopril 6.25 mg test dose and Caps Trandolapril 0.5mg or 1.0mg or 2.0 mg (depending on symptoms ie. hypotension)
Drug: Captopril Test Dose and Trandolapril — Caps Captopril 6.25 mg test dose and Caps Trandolapril 0.5mg or 1.0mg or 2.0 mg (depending on symptoms ie. hypotension)

SUMMARY:
Abundant evidence suggests that Angiotensin Converting Enzyme (ACE) inhibition potentially could reduce the hazardous effects of aortic stenosis and improve haemodynamics. The treatment seems safe even in patients with severe stenosis. There are however no randomised clinical trials that can confirm this hypothesis.

DETAILED DESCRIPTION:
Traditionally vasodilators are contraindicated in patients with aortic stenosis. Although no controlled data exists it is believed to be hazardous to reduce afterload, including treatment with angiotensin converting enzyme (ACE) inhibitors, in these patients with aortic stenosis due to the risk of increased transaortic gradient and thus severe hypotension and myocardial hypoperfusion. There is now growing evidence both experimental and clinical that ACE inhibition could have beneficial effects on left ventricular hypertrophy, diastolic function, acute, and possibly chronic haemodynamic parameters in patients with aortic stenosis.

There is, however, a lack of clinical randomized trials that could confirm these findings.

Aims

Prospective double blinded randomised study investigating the safety and effects of treatment with ACE-inhibitor in patients with severe aortic stenosis. Effects will be measured on :

* Invasive measured haemodynamic parameters (Swann-Ganz)
* Working capacity
* Diastolic and systolic function (measured with tissue Doppler echocardiography)
* Blood pressure
* B-type natriuretic peptide (BNP)

Patients

32 patients with symptomatic aorta stenosis recruited from Rigshospitalet department of cardiology. Patients referred for evaluation prior to surgical intervention with insertion of a valvular prosthesis will be screened.

Additional 32 patients with asymptomatic aorta stenosis will be recruited from Rigshospitalet and other cardiology departments.

Methods

Recruitment

Patients with symptomatic severe aortic stenosis scheduled for aortic valve replacement at The Heart Centre at Rigshospitalets department of cardiology will be recruited.

Patients with severe asymptomatic aortic stenosis on Rigshospitalet will be recruited. If it is necessary, patients from other hospitals will be recruited.

Randomisation

After baseline screening, patients will be randomized to active treatment or placebo. Half of the patients will have ACE-inhibitors (Captopril-test dose after this Trandolapril) the other half placebo.

Administration of medicine

ACE-inhibitor/placebo administration will be double blinded and performed by a hospital pharmacist not involved in any other part of the project.

All patients will be hospitalised in the intensive care unit for the first 3 days to evaluate the acute haemodynamic changes when they start the treatment. If the patients have no symptoms after the 3 days they will discharge for further treatment for up to 8 weeks. Visits are planned after 2 and 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Valvular aortic stenosis with a aortic valve area < 1, 0 cm2
* Age > 18 years
* Willingness to give written informed consent
* For patients with symptomatic aortic stenosis at least one of following:

  * Stable angina pectoris
  * Syncope at exertion
  * Dizziness at exertion
  * Previous pulmonary oedema
  * Patients in New York Heart Association functional class II-IV

Exclusion Criteria:

* Sitting systolic pressure < 100 mmHg
* Creatinine > 200 mM at screening
* Renal artery stenosis
* Pregnancy or planned pregnancy
* Participation in other studies
* Any patient characteristic that may interfere with compliance with the study protocol
* Treated with ACE-inhibitor or angiotensin receptor blocker within the last month
* Known allergy to ACE-inhibitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2005-11; Study Completion 2008-10 (Estimated)

PRIMARY OUTCOMES:
Treatment with ACE-inhibitors improves haemodynamic parameters in patients with severe aortic stenosis. | 8 weeks

SECONDARY OUTCOMES:
Treatment with ACE-inhibitors: | 8 weeks
Increases working capacity in patients with severe aorta stenosis. | 8 weeks
Improves systolic and diastolic function on left ventricle. | 8 weeks
In patients with severe aortic stenosis is safe. | 8 weeks
Degrease wall stress in left ventricle. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Morten Dalsgaard, MD, Principal Investigator — Rigshospitalet, Denmark; Christian Hassager, MD, Phd, Principal Investigator — Rigshospitalet, Denmark; Peter Clemmensen, MD, Phd, Principal Investigator — Rigshospitalet, Denmark; Peer Grande, MD, Phd, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen University Hospital, Copenhagen, KBH Ø, Denmark

REFERENCES:
- [Background] Routledge HC, Townend JN. ACE inhibition in aortic stenosis: dangerous medicine or golden opportunity? J Hum Hypertens. 2001 Oct;15(10):659-67. doi: 10.1038/sj.jhh.1001260. PMID 11607794
- [Derived] Dalsgaard M, Kjaergaard J, Pecini R, Iversen KK, Kober L, Moller JE, Grande P, Clemmensen P, Hassager C. Predictors of exercise capacity and symptoms in severe aortic stenosis. Eur J Echocardiogr. 2010 Jul;11(6):482-7. doi: 10.1093/ejechocard/jeq002. Epub 2010 Feb 6. PMID 20139439